CLINICAL TRIAL: NCT06157762
Title: Comparison of the Effectiveness of Preoperative Ultrasound-Guided Erector Spine Plane Block and Erector Spine Plane Block Performed by the Intraoperative Surgeon in Postoperative Analgesia in Patients Undergoing Lumbar Disc Herniation Surgery
Brief Title: Open Technique Erector Spinae Plane Block in Spinal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Gökçe Gişi, Assistant Professor, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022/26-05
Record Dates: First submitted 2023-11-27; First posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Postoperative Pain; Erector Spinae Plane Block in Spinal Surgery
Keywords: Pain; postoperative analgesia; Erector spinae plane block; Spinal surgery; Open Technique
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESPB performed by surgeon (Experimental): The transverse process of the vertebra will be observed by the surgeon intraoperatively. Local anesthetic medication will be applied between the transverse process and the ESP muscle group.
  Interventions: Procedure: Erector spinae plane block performed by surgeon
- Erector spinae plane block (Active Comparator): The ultrasound-guided erector spinae plane block will be applied preoperatively.
  Interventions: Procedure: Erector spinae plane block

INTERVENTIONS:
Procedure: Erector spinae plane block — ultrasound guided lumbar erector spinae plane block
  Arms: Erector spinae plane block
Procedure: Erector spinae plane block performed by surgeon — Erector spinae plane block performed by surgeon
  Arms: ESPB performed by surgeon

SUMMARY:
Erector spinae plane (ESP) block is an interfacial plane block with visceral and somatic analgesic activity at paraspinal muscles.ESPB has been successfully applied as a part of multimodal analgesia in treating postoperative pain in spinal surgery. However, it may be difficult or impossible to perform lumbar ESPB in obese patients or cases of increased lumbar lordosis. This study aims to investigate the effectiveness of ESPB applied by the intraoperative surgeon.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III patients
* Agreed to participate in the study

Exclusion Criteria:

* Patients with infection at the injection site
* Coagulopathy Allergy to amide-type local anesthetics
* History of peripheral neuropathy
* Hepatic and/or renal failure
* Refusing the procedure
* Patients with heart disease
* Patients who have previously undergone surgery from the same area

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
opioid consumption | up to 24 hour
  The amount of morphine consumed in milligrams in the first 24 hours was determined with a patient-controlled analgesia pump.